CLINICAL TRIAL: NCT00100893
Title: A Phase I Prevention Trial of ACTIVIN Grape Seed Extract as an Aromatase Inhibitor In Healthy Postmenopausal Women at Risk for Breast Cancer
Brief Title: IH636 Grape Seed Extract in Preventing Breast Cancer in Postmenopausal Women at Risk of Developing Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 03178; P30CA033572 (NIH); CHNMC-IRB-03178; CDR0000407637 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2005-01-06; First posted 2005-01-07 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Grape Seed Proanthocyanidins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dietary Supplement: grape seed proanthocyanidin extract (Experimental): Administered orally.
  Interventions: Dietary Supplement: IH636 grape seed proanthocyanidin extract

INTERVENTIONS:
Dietary Supplement: IH636 grape seed proanthocyanidin extract — Dose escalation as follows: 50 mg/day, 300 mg/day, 1000 mg/day, 2000 mg/day, 2800 mg/day, 4000 mg/day, 4800 mg/day and 6000 mg/day in separate patient groups for each dosage

SUMMARY:
RATIONALE: Chemoprevention is the use of certain drugs to keep cancer from forming, growing, or coming back. The use of IH636 grape seed extract may prevent breast cancer.

PURPOSE: This phase I trial is studying the side effects and best dose of IH636 grape seed extract in preventing breast cancer in postmenopausal women at risk of developing breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of IH636 grape seed proanthocyanidin extract, in terms of suppression of estrogen biosynthesis, in healthy post-menopausal women at high risk of developing breast cancer.
* Determine the safety and tolerability of this dietary supplement, in terms of symptoms and changes in markers of bone and lipid metabolism and in markers of nonspecific adrenal suppression, in these participants.
* Determine, preliminarily, an optimum biologic dose of this dietary supplement, as defined by suppression of serum estradiol, in these participants.
* Determine a minimum duration of use of this dietary supplement to achieve aromatase inhibition in these participants.

OUTLINE: This is a pilot, dose-finding, placebo-controlled study.

Participants receive oral placebo once or twice daily on days -14 to 0. Participants then receive oral IH636 grape seed proanthocyanidin extract once or twice daily on days 1-85. Treatment continues in the absence of toxicity.

Cohorts of 6 participants receive one of four dose levels of IH636 grape seed proanthocyanidin extract up to an established safe dose.

PROJECTED ACCRUAL: A total of 24 participants will be accrued for this study within 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* At risk of developing breast cancer
* No history of breast cancer or ductal carcinoma in situ

PATIENT CHARACTERISTICS:

Age

* 40 to 75

Sex

* Female

Menopausal status

* Postmenopausal, defined by 1 of the following criteria:

  * No spontaneous menses for ≥ 12 months
  * Prior bilateral oophorectomy
  * Prior hysterectomy with follicle-stimulating hormone within menopausal range

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Hemoglobin ≥ 9.0 g/dL
* Platelet count ≥ 100,000/mm^3
* WBC ≥ 3,500/mm^3
* Absolute granulocyte count ≥ 1,500/mm^3
* No coagulation disorders

Hepatic

* SGOT and SGPT ≤ 2 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN

Renal

* Creatinine ≤ 1.5 times ULN

Cardiovascular

* No major illness of the cardiovascular system

Pulmonary

* No major illness of the respiratory system

Other

* No history of other invasive cancer within the past 5 years except squamous cell or basal cell skin cancer
* No major systemic infection
* No Cushing's syndrome or adrenal insufficiency
* No osteoporosis, defined as a bone mineral density T-score ≥ -2.5 on dual-energy x-ray absorptiometry scan (calcium and/or cholecalciferol [vitamin D] supplementation AND/OR bisphosphonate therapy allowed provided participant is on a stable dose during study participation)

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* More than 3 months since prior hormone-modifying medications, including any of the following:

  * Oral contraceptives
  * Hormone replacement therapy
  * Selective estrogen receptor modifiers
  * Aromatase inhibitors
  * Gonadotropin-releasing hormone modifiers
* Concurrent dehydroepiandrosterone (DHEA) allowed, provided dose remains constant during study participation

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* No red wine, red grapes, or white button mushrooms directly before or during study treatment

  * White and seedless grapes allowed
* No other concurrent therapy

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2005-01; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Estrogen suppression as measured by serum estradiol, estrone, estrone sulfate, and sex hormone binding globulin | at 1, 2, 4, 8, and 12 weeks

SECONDARY OUTCOMES:
Androgenic effects as measured by serum testosterone, androstenedione, dehydroepiandrosterone (DHEA), and dehydroepiandrosterone sulfate (DHEAS) | at 1, 2, 4, 8, and 12 weeks
Lipid effects as measured by total cholesterol, LDL, HDL, and triglycerides | at 12 weeks
Bone metabolic effects as measured by bone-specific alkaline phosphatase and N-telopeptides | at 12 weeks
Insulin regulatory effects as measured by insulin-like growth factor 1 (IGF1) and insulin-like growth factor-binding protein 3 (IGFBP3) | at 12 weeks
Pharmacokinetics as measured by procyanidins | before and after first dose and then at 1, 2, 4, 8, and 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- City of Hope Comprehensive Cancer Center, Duarte, California, United States